CLINICAL TRIAL: NCT01613300
Title: Ofatumumab as Part of the Reduced Intensity Conditioning Regimen (RIC) for Patients With High Risk B Non Hodgkin's Lymphoma Undergoing Allogeneic Hematopoietic Cell Transplantation
Brief Title: Study of OFATUMUMAB as Part of the Scheme of Reduced Intensity Conditioning in High Risk Non-Hodgkin Lymphoma B Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Español de Linfomas y Transplante Autólogo de Médula Ósea (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GELTAMO-O-CRT-2011; 2011-004729-29 (EudraCT Number)
Record Dates: First submitted 2012-06-05; First posted 2012-06-07 (Estimated); Last update posted 2021-05-26 (Actual); Status verified 2021-01

CONDITIONS: B-Cell Lymphomas
Keywords: hodgkin; disease; ofatumumab
MeSH Terms: conditions — Lymphoma, B-Cell; Disease | interventions — ofatumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ofatumumab (Experimental): Ofatumumab as part of the reduced intensity conditioning regimen (RIC)
  Interventions: Drug: Ofatumumab

INTERVENTIONS:
Drug: Ofatumumab — Ofatumumab as part of the reduced intensity conditioning regimen (RIC)
  Other Names: ARZERRA

SUMMARY:
The aim of this study is rate of acute graft-versus-host disease II-IV measured at day +365according to conventional criteria (Przepiorka et al. 1995) in patients with high risk non-Hodgkin lymphoma B subjects with Allogeneic Stem Cell Transplant

DETAILED DESCRIPTION:
In addition to above:

* Rate of progression-free survival (PFS) at 12, 24, 36 and 60 months post-transplant defined as the time between the infusion of progenitors and the disease progression or death. Patients alive or in complete remission will be censored at the time of last follow up
* Transplant-related mortality (TRM) at 12, 24, 36 and 60 months after transplantation, defined as any death not caused directly by lymphoma (any death caused by complications related to transplantation).
* Overall survival (OS) defined as the time between infusion of progenitors and the patient's death from any cause. Alive Patients will be censored at the time of last follow-up
* Incidence of chronic graft versus host disease (GVHD) wide at 1 and 5 years according to conventional criteria (Atkinson et al. 1989) and Filipovich et al. (BBMT, 2005).
* Rate of event-free survival (DFS) defined as time interval between diagnosis of lymphoma and lymphoma progression or relapse or death if the above does not occur.
* Successful graft implantation: is defined as:

  1. º: three consecutive days with absolute neutrophil count greater than 0.5 * 109 / L
  2. ° thrombocythemia exceeds 20 * 109 / L.
* Reconstitution of the immune system: lymphocyte count populations CD20, CD3, CD4 and CD8 and immunoglobulinemia serum (days +100, 180, 360, 18 months and 24 months).
* intercurrent infections. All sorts of infections (viral, fungal and bacterial)will be recorded
* Safety assessment by the standards of Common Terminology Criteria for adverse events v. 4.0

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who have given their informed consent before any study-specific procedures
2. Histopathological diagnostic of NHL cell B CD 20 + B of different histologic subtypes:
3. High risk CD +20 Lymphoma having at least one of the following characteristics:

   * Less than a partial remission after two courses of treatment
   * Relapse after autologous peripheral blood stem cell (PBSCT)
   * Evidence of measurable disease (With CT and PET or PET / CT) three months after PBSCT
   * Hematopoietic precursors improper count in patients with relapsed or partial remission after two treatment lines that prevent the realization of a PBSCT.
   * Patients after first relapse in RP after two lines of treatment in whom the probability of freedom from progression per year is very low due to risk factors such as: first CR less than 12 months after PBSCT low SLP, etc..
4. Age between 18 and 65 years
5. ECOG between 0 to 1 (Appendix III).
6. Subjects who are HBgAG negative, anti-HBc positive and HBV DNA negative may be include in the study but must undergo HBV DNA monitoring
7. Adequate lung Function
8. Cardiac ejection greater than 40% as measured by scintigraphy or echocardiography.
9. Adequate renal and hepatic function defined by the following biochemical parameters
10. The disease status prior to transplantation had to be in place in accordance with the criteria of Revised Response Criteria for Malignant Lymphoma, Cheson 2007. CT and PET or PET / CT.
11. Availability of a histocompatible donor (9 to 10/10 loci) family or unrelated
12. Adults with ability to procreate must commit to use an effective method of birth control during the study treatment and at least 6 months.

Exclusion Criteria:

1. Refractory disease at the time of transplantation
2. Progressive disease at the time of transplantation.
3. ECOG≤2
4. Lymphoma associated with infection with human immunodeficiency virus (HIV).
5. Test positive for HIV.
6. Presence of anti-murine antibodies (HAMA) or (HACA).
7. Treatment with any marketed or experimental drug administered not in a period between 5 terminal half-lives of clearance of therapy or 4 weeks before enrollment
8. Participation in another interventional clinical trial.
9. Prior treatment with anti-CD20 monoclonal antibody or alemtuzumab within 3 months prior to start of therapy. This is generally required and may be excluded as applicable.
10. Hepatitis B positive serology
11. Positive serology for Hepatitis B (HB) defined as a positive test for HBsAg.
12. Positive serology for hepatitis C (HC) defined as a positive test for HCAb.
13. Active liver or biliary disease (with exception of Gilbert's disease, cholelithiasis, metastases).
14. Other past or current malignancy.
15. Chronic infectious disease that requires ongoing treatment with systemic antibiotics, antifungal or antiviral drugs
16. History of cerebrovascular disease active in the last 6 months or event with significant symptoms or sequelae.
17. Clinically significant heart disease, such as unstable angina, acute myocardial infarction in the six months prior to inclusion, congestive heart failure (grades III-IV NYHA) and arrhythmia unless it is controlled by treatment, except for premature or disorders Mild driving.
18. Concurrent medical disorder, uncontrolled and important, such as kidney disease, liver, digestive, endocrine, pulmonary, neurological, brain, psychiatric, or which in the opinion of the investigator may represent a risk to the patient
19. Pregnancy or breastfeeding
20. Women of childbearing potential, including those whose last menstrual period was one year prior to screening.
21. Men unable or unwilling to use contraception
22. Patients with hypersensitivity to fludarabine, melphalan, thiotepa, tacrolimus, sirolimus and / or any excipients.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2012-04-04 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Rate of acute grade II-IV graft-versus-host disease at 1 year | 5 years follow-up
  According to conventional criteria. This endpoint will be descriptively reported. Confidence intervals (95% bounds) will be provided. The rate will be analyzed in all patients enrolled at the clinical trial and that no major violation has been produced.

SECONDARY OUTCOMES:
To analyze the complete response rate after treatment. Further secondary outcomes as described in study summary | 5 years follow up
  To analyze the complete response rate after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Maria Dolores Caballero, MD, Principal Investigator — Hospital Clinico de Salamanca
Locations (10):
- Spain (10):
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Reina Sofia, Córdoba
  - H.U. 12 de Octubre,, Madrid
  - H.U. Gregorio Marañón,, Madrid
  - H.U. La Paz, Madrid
  - Complejo Hospitalario Carlos Haya, Málaga
  - H. Morales Meseguer., Murcia
  - H. Clinico de Salamanca, Salamanca
  - Hospital Virgen del Rocío, Seville
  - H. La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cabrero M, Lopez-Corral L, Jarque I, de la Cruz-Vicente F, Perez-Lopez E, Valcarcel D, Sanz J, Espigado I, Orti G, Martin-Calvo C, de la Serna J, Caballero D; Grupo Espanol de Trasplante Hematopoyetico (GETH) and Grupo Espanol de Linfomas y Trasplante Autologo (GELTAMO). Ofatumumab as part of reduced intensity conditioning in high risk B-cell lymphoma patients: final long-term analysis from a prospective multicenter Phase-II Trial. Bone Marrow Transplant. 2024 Mar;59(3):359-365. doi: 10.1038/s41409-023-02171-5. Epub 2024 Jan 2. PMID 38167647